CLINICAL TRIAL: NCT03723512
Title: Sub-project of the Clinical Protocol ACH471-205 "An Open-Label Phase 2 Proof-of-Concept Study in Patients With C3 Glomerulopathy (C3G) or Immune-Complex Membranoproliferative Glomerulonephritis (IC-MPGN) Treated With ACH-0144471"
Brief Title: Non-contrast Enhanced MRI in Patients With C3 Glomerulopathy (C3G) or Immune-complex Membranoproliferative Glomerulonephritis (IC-MPGN) Enrolled in the ACH471-205 Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Subproject MRI ACH471-205
Record Dates: First submitted 2018-10-22; First posted 2018-10-29 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: C3 Glomerulonephritis; C3 Glomerulopathy; Immune Complex Membranoproliferative Glomerulonephritis; IC-MPGN; Dense Deposit Disease
Keywords: Non-contrast enhanced MRI; Diffusivity; Renal microstructure; Renal function; C3G; IC-MPGN
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole group (Experimental): Whole group
  Interventions: Device: Non contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Device: Non contrast-enhanced magnetic resonance imaging — Non contrast-enhanced magnetic resonance imaging

SUMMARY:
Functional and quantitative renal magnetic resonance imaging (MRI) has seen a number of recent advances, and techniques are now available that can generate quantitative imaging biomarkers with the potential to improve the management of kidney disease.

However, there are knowledge gaps that must be addressed before renal MRI methods could be more widely adopted in clinical research and ultimately be transferred to clinical practice, including the biological basis of different MRI biomarkers, and how the application of these biomarkers will improve patient care.

Among renal MRI techniques, renal diffusion weighted MRI (DWI) has been increasingly used in the last decade, showing high potential as a surrogate and monitoring biomarker for interstitial fibrosis in chronic kidney disease (CKD), as well as a surrogate biomarker for the inflammation in acute kidney diseases that may impact patient selection for renal biopsy in acute graft rejection.

Within the ready-to-start ACH471-205 clinical trial, an Open-Label Phase 2 Proof-of-Concept Study in Patients with C3 Glomerulopathy (C3G) or Immune-Complex Membranoproliferative Glomerulonephritis (IC-MPGN) treated with ACH-0144471, aimed at evaluating the efficacy of 12 months of oral ACH-0144471 in patients with C3G or IC-MPGN, patients will undergo baseline and 12-month follow-up renal biopsies, and renal function will be assessed over time by estimated or measured (when available) glomerular filtration rate (GFR). Adding multi-parametric NCE-MRI to the examinations under the ACH471-205 study protocol will give the opportunity to elucidate, in a well-defined cohort of patients, the potential of NCE-MRI as biomarker of renal microstructure and functional change.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of C3G or IC-MPGN;
* Patients enrolled in the ACH471-205 study at the Bergamo center;
* No contraindications to perform MRI.

Exclusion Criteria:

- Ferro-magnetic prosthesis, aneurysm clips, severe claustrophobia or other contraindications or exclusions interfering with the MRI assessment.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Median diffusivity (D) in the kidney, renal cortex and medulla. | At baseline (prior to baseline biopsy).
Median diffusivity (D) in the kidney, renal cortex and medulla. | At 12 months (prior to follow-up biopsy).

SECONDARY OUTCOMES:
Renal artery blood flow and renal plasma flow. | At baseline (prior to baseline biopsy).
Renal artery blood flow and renal plasma flow. | At 12 months (prior to follow-up biopsy).
Change in median diffusivity in the kidney, renal cortex and medulla after 12-month treatment with ACH-0144471. | At 12 months follow-up.
Change in renal artery blood flow and renal plasma flow after 12-month treatment with ACH-0144471. | At 12 months follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro di Ricerche Cliniche per le Malattie Rare Aldo e Cele Daccò, Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Selby NM, Blankestijn PJ, Boor P, Combe C, Eckardt KU, Eikefjord E, Garcia-Fernandez N, Golay X, Gordon I, Grenier N, Hockings PD, Jensen JD, Joles JA, Kalra PA, Kramer BK, Mark PB, Mendichovszky IA, Nikolic O, Odudu A, Ong ACM, Ortiz A, Pruijm M, Remuzzi G, Rorvik J, de Seigneux S, Simms RJ, Slatinska J, Summers P, Taal MW, Thoeny HC, Vallee JP, Wolf M, Caroli A, Sourbron S. Magnetic resonance imaging biomarkers for chronic kidney disease: a position paper from the European Cooperation in Science and Technology Action PARENCHIMA. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii4-ii14. doi: 10.1093/ndt/gfy152. PMID 30137584
- [Background] Caroli A, Schneider M, Friedli I, Ljimani A, De Seigneux S, Boor P, Gullapudi L, Kazmi I, Mendichovszky IA, Notohamiprodjo M, Selby NM, Thoeny HC, Grenier N, Vallee JP. Diffusion-weighted magnetic resonance imaging to assess diffuse renal pathology: a systematic review and statement paper. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii29-ii40. doi: 10.1093/ndt/gfy163. PMID 30137580
- [Derived] Villa G, Daina E, Brambilla P, Gamba S, Leone VF, Carrara C, Rizzo P, Noris M, Remuzzi G, Remuzzi A, Caroli A. Functional Magnetic Resonance Imaging to Monitor Disease Progression: A Prospective Study in Patients with Primary Membranoproliferative Glomerulonephritis. Nephron. 2024;148(6):367-378. doi: 10.1159/000534893. Epub 2023 Nov 3. PMID 37926085